CLINICAL TRIAL: NCT01230411
Title: A Double-blind, Placebo-controlled Pilot Study to Collect and Evaluate Data on the Use of Intravenous Ibuprofen in the Treatment of an Acute Migraine Attack
Brief Title: Pilot Study to Collect and Evaluate Data on the Use of IV* Ibuprofen in the Treatment of an Acute Migraine Attack
Acronym: intravenous
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SDS/IVIb/01
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Results first posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Episodic Migraine
Keywords: Episodic migraine
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): IV saline administration as placebo
  Interventions: Other: saline placebo
- Ibuprofen (Experimental): IV ibuprofen
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Other: saline placebo — 250 cc of placebo administered IV
  Arms: placebo
Drug: Ibuprofen — 800 mg ibuprofen in 250 cc saline administered IV
  Other Names: Caldolor
  Arms: Ibuprofen

SUMMARY:
This is a pilot trial to collect data on the use of intravenous ibuprofen (IVIb) in the treatment of an acute migraine attack. Data will be collected on the efficacy of IVIb in subjects who are treated with study medication between 2 and 72 hours from time of onset of headache.

Periodic safety and efficacy assessments will be performed prior to and after study drug administration.

Null hypothesis: There is no difference in the proportion of subjects in the 2 treatment groups (active treatment and placebo) who have pain relief at 2 hours after the completion of the double-blind treatment infusion. Pain relief is defined as a reduction in headache pain level from severe or moderate decreased to mild or headache-free, respectively.

DETAILED DESCRIPTION:
This is a 3 visit trial: screening visit, treatment visit, and final visit. Screening visit and a treatment visit may occur on the same day. Additionally, there will be one follow-up phone call at 24 hours post-dose. Subjects will be screened and the investigator will determine whether or not the subject experiences episodic migraine headaches. When a potential subject is seen as an office patient at the Jefferson Headache Center, has a headache, and is referred by the PI or co-investigator to this study, the referring study physician will document that the subject's cognition is intact and the subject is able to understand and sign the informed consent at that time. If the potential subject's cognition is affected by the migraine, the subject must return to the Jefferson Headache Center for the research screening visit when the headache and cognitive difficulties have resolved. Subjects who are not being seen as an office patient on the day of screening must be headache-free at the time of screening.

Those subjects who meet the qualifying criteria will be eligible for treatment in the study. Subjects who qualify will be asked to come to the Jefferson Headache Center within 2 to 72 hours following the onset of pain.

IVIb or placebo will be administered intravenously as the study treatment. For active treatment, 800 mg of injectable ibuprofen will be placed in 250 ml of normal saline, and infused over 7-10 minutes. (Infusion time may be increased up to 1 hour if necessary due to possible anatomical restrictions). The placebo group will receive 250 ml of normal saline, infused over 7-10 minutes. (Infusion time may be increased up to 1 hour if necessary due to possible anatomical restrictions). Safety and efficacy assessments will be made periodically just prior to and after administration of study drug. Migraine pain and associated symptom assessments will be measured by the subjects for 24 hours from the administration of study drug for the treated attack. If subjects still have a moderate to severe headache at 2 hours after receiving double-blind study drug, they will receive a rescue dose of 800 mg. IV Ibuprofen. Subjects will be discharged at 4 hours post study drug dose, or when clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 18 and 65, inclusive
* Subject diagnosed with episodic migraine, with or without aura according to ICHD-2 criteria for at least one-year prior to screening
* Subject experiences between 2-10 migraine attacks per month (during the previous 6 months) with no more than 15 days of headache per month.
* Subject is using or agrees to use for the duration of participation a medically acceptable form of contraception (as determined by investigator), if female and of child-bearing potential
* Subject is able to come for 4 hour in-clinic treatment of an acute migraine attack
* Subjects are able to understand and comply with all study procedures.
* Subject provides written informed consent prior to any screening procedures being conducted
* If subject is on an allowable migraine preventive medication, the dose has been stable for at least 4 weeks prior to screening and the dose will remain stable throughout study participation.

Exclusion Criteria:

* Unable to make a reliable self-report of pain intensity to pain relief
* Use of analgesic or opioid within 24 hours of onset of headache to be treated with study medication. (If subject has an eligible headache and has taken a triptan or DHE within 24 hours, but greater than 2 hours before study drug dosing, they can be treated with study medication.)
* Patients taking the following medications on a regular basis: warfarin, lithium, ACE-inhibitors, loop diuretics, thiazide diuretics, ARBs, and methotrexate.
* Patients with active, clinically significant anemia
* Patients with a history or evidence of asthma
* Patients with a history heart failure
* Subjects with severely impaired hepatic or renal function, as determined by the investigator
* Patients with a history of allergy or hypersensitivity to any component of IVIb, aspirin (or aspirin related products), NSAIDs, or COX-2 inhibitors
* Pregnant or nursing women
* Patients who have a history of congenital bleeding diathesis (e.g., hemophilia) or any active clinically significant bleeding, or have underlying platelet dysfunction including (but not limited to) idiopathic thrombocytopenic purpura, disseminated intravascular coagulation, or congenital platelet dysfunction
* Patients who have GI bleeding that required medical intervention within the previous 6 weeks (unless definitive surgery has been performed.)
* Patients who have a platelet count less than 100,000, as determined within the 28 days prior to treatment
* Pre-existing or current dependence on opioids.
* Subjects who have participated in an investigational drug trial in the 30 days prior to the screening visit
* Subjects with uncontrolled hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-06; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D. Silberstein, M.D., Principal Investigator — Jefferson Headache Center
Locations (1):
- Jefferson Headache Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Yuan H, Curran JG, Keith SW, Hopkins MM, Silberstein SD. Intravenous ibuprofen for acute treatment of migraine: A double-blind, randomized, placebo-controlled pilot study. Headache. 2021 Oct;61(9):1432-1440. doi: 10.1111/head.14214. Epub 2021 Oct 3. PMID 34601736

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Ibuprofen
Started | 21 | 23
Completed | 21 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ibuprofen | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (12.1) | 42.8 (10.5) | 41.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 4 | 7 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Migraine Duration Since onset (years) [Mean (Standard Deviation); unit: years] | 16.4 (10.4) | 23.6 (11.4) | 20 (10.9)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Proportion of Subjects in Control and Active Treatment Groups Who Have Pain Relief at 2 Hours After the Completion of the Double-blind Treatment Infusion.
Description: Comparison of proportion of subjects in each treatment group (active treatment and placebo) who have pain relief at 2 hours after the completion of the double-blind treatment infusion. Pain relief is defined as a reduction in headache pain level from severe or moderate decreased to mild or headache-free, respectively.
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ibuprofen
Number analyzed (Participants) | 21 | 23
Participants | 10 | 17
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen; Test type: Superiority; p = 0.078, Regression, Logistic; Odds Ratio (OR) = 3.12, 95% CI 2-sided [0.88 to 11.0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of treatment ( which could take up to 1 hr), then at post treatment time points: 30 min , 1hour, 2 hour as well as during the 24 hr post treatment phone call and at 1 week follow up.
Arm/Group | Placebo | Ibuprofen
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23
Other Adverse Events (participants affected / at risk) | 3/21 | 4/23
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | Ibuprofen (N=23)
arm pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Gastrointestinal disturbance (Gastrointestinal disorders) | 2 | 0
dizziness (Nervous system disorders) | 0 | 1
Cold sensitivity (Nervous system disorders) | 0 | 1
Neck pain (Nervous system disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Slow enrollment and small sample size impacted the type 1 error, study power, and quality. The randomization failed to balance the distribution of migraine duration between the two groups. No blinding assessment was done. The primary endpoint of 2HR pain relief for acute migraine treatment was the most common outcome measure at the time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-07-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT01230411/Prot_SAP_000.pdf
  • Informed Consent Form (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT01230411/ICF_001.pdf